CLINICAL TRIAL: NCT06804369
Title: Benchmarking and Mechanisms of Change During Intensive Psychodynamic Therapy for Personality Disorders: A Naturalistic Process-Outcome Study
Brief Title: Benchmarking and Change Mechanisms in Personality Disorder Treatment
Status: Active, not recruiting | Type: Observational
Sponsor: KU Leuven (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Celine De Meulemeester, Dr., KU Leuven
Other Study IDs: S67356
Record Dates: First submitted 2025-01-21; First posted 2025-02-03 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Personality Disorders
Keywords: personality disorders; change mechanisms; benchmarking; epistemic trust; mentalizing; resilience; psychodynamic therapy
MeSH Terms: conditions — Personality Disorders | interventions — Psychotherapy, Psychodynamic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Personality Disorder Patients: All patients consecutively admitted to the KLIPP treatment unit (UPC KU Leuven, Belgium) until the target sample size (N = 110) is reached. All patients have been referred to this specialized treatment because of prominent personality disorder pathology and undergo multidisciplinary assessment by a psychiatrist, clinical psychologist and social worker.
  Interventions: Behavioral: Intensive psychodynamic therapy (PDT)

INTERVENTIONS:
Behavioral: Intensive psychodynamic therapy (PDT) — The KLIPP treatment unit (UPC KU Leuven, campus Kortenberg) provides intensive psychodynamic treatment (PDT) for patients with different types of PDs. There are three different programs that differ in treatment intensity: (1) inpatient treatment program (5 days a week), (2) day treatment program (4 days a week), and (3) a part-time outpatient treatment program of two half days per week. Patients attend one of these programs and stay in the program for at least 6 months (with an average duration of 8 months). The programs include individual and group psychodynamic psychotherapy as well as art, music and psychomotor therapy.
  Other Names: Psychodynamic Psychotherapy

SUMMARY:
Personality disorders (PDs) are severe mental disorders characterized by pathological personality traits as well as problems in identity and interpersonal relationships (American Psychiatric Association, 2013). Several effective psychotherapies for PDs have been developed in the past decades, however, two important questions regarding PD treatment have not been sufficiently addressed: (1) how effective are PD treatments outside of the controlled settings of randomized controlled trials (RCTs); (2) are the effects of PDT clinically meaningful; and (3) what are the core processes that produce change in PD treatment? The present observational study aims to address these research gaps by (1) comparing the effects of intensive psychodynamic therapy (PDT) for PDs in a naturalistic setting to benchmarks found in RCTs; (2) analyzing which proportion of patients achieves clinically meaningful change and (3) investigating whether outcomes in intensive PDT are associated with a number of theoretically expected mechanisms of change.

DETAILED DESCRIPTION:
Personality disorders (PDs) are characterized by problems with identity and interpersonal relationships and the presence of pathological personality traits (American Psychiatric Association, 2013). Personality disorders are prevalent, affecting about 6 - 9.5% of people in the community (Winsper et al., 2020) and result in increased morbidity and mortality (Grant et al., 2008). Several effective psychotherapies for PDs have been developed in the past decades. Meta-analyses of randomized controlled trials (RCTs) demonstrate that psychotherapy for PDs is efficacious and that different treatment models for PDs produce comparable effects (Budge et al., 2013; Cristea et al., 2017; Storebø et al., 2020). However, two important questions remain: (1) how effective are PD treatments outside of the controlled settings of RCTs and (2) what are the core processes that produce change in PD treatment?

First, evidence on the efficacy of PD treatment in controlled circumstances (RCTs) does not necessarily translate directly to the effectiveness of treatment as it is actually being delivered in routine clinical practice. Several studies have demonstrated the effectiveness of PD treatment in naturalistic settings (Gregory & Sachdeva, 2016; Lowyck et al., 2015), however, these studies have not systematically compared their effects with those from published RCTs (Malmivaara, 2015). Therefore, the primary aim of the present study is to compare the effects of intensive psychodynamic therapy (PDT) for PDs in a naturalistic setting to benchmarks found in RCTs. Specifically, the primary objective of this study is to investigate the non-inferiority with a margin of d = 0.2 of intensive PDT for PDs as it is delivered in routine clinical practice compared to benchmarks from published RCTs of PDT for PDs. The benchmarks are created by meta-analytically aggregating the effects found in well-conducted RCTs following the methods proposed by Minami et al. (2008). The primary outcome is change in general symptom severity as measured by the global severity index (GSI) on the Brief Symptom Inventory (BSI) from start to end of treatment (approximately 8 months after the start of treatment).

Second, the effectiveness of intensive PDT for PD in terms of pre-post effect sizes will be investigated as well as clinical significant change (CSC) and deterioration using reliable change indices (Jacobson & Truax, 1991) from baseline to treatment termination as well as 6-month and 1- and 2-year follow up, on the following outcomes: psychological distress (Brief Symptom Inventory; BSI), borderline personality disorder symptoms (Personality Assessment Inventory for BPD; PAI-BOR); personality functioning (Level of Personality Functioning Scale; LPFS), interpersonal functioning (Inventory of Interpersonal Problems; IIP), post-traumatic stress (Post-traumatic stress disorder Checklist for DSM-5; PCL-5), resilience (Connor-Davidson Resilience Scale; CD-RISC) and quality of life (EQ-5D).

Third, in order to ensure that existing therapies for PDs focus on the actual core processes that produce change, more research is needed to address why and how treatment for PD works (Kramer, 2018). The present study's secondary aim is therefore to investigate whether outcomes in intensive PDT are associated with a number of theoretically expected mechanisms of change. It has been argued that successful treatment for PDs fosters epistemic trust, that is, trust in communicated knowledge, which in turn allows for the re-emergence of learning from benign social influences, increasing resilience and reducing PD symptoms (Fonagy et al., 2019). Epistemic trust is thus theoretically considered a core change mechanism in all effective treatments for PD, however, no study to date has empirically tested this. The secondary objective of the present study is to investigate whether trajectories of change in epistemic trust, mistrust and credulity across treatment (as measured using the Epistemic Trust, Mistrust and Credulity Questionnaire, ETMCQ) are associated with the trajectories of symptom change across treatment (as measured using the Brief Symptom Inventory, BSI, and the Personality Assessment Inventory for borderline PD, PAI-BOR) using parallel process growth curve modeling (MacCallum et al., 1997). Mentalizing and therapeutic alliance are investigated as secondary change mechanisms to assess the relative importance of epistemic trust as a change mechanism in the treatment of PD.

This observational clinical study aims to recruit N = 110 PD patients consecutively admitted to a treatment unit that specializes in intensive PDT for PDs (Klipp, UPC KU Leuven, Belgium). Patients follow one of three programs that differ in treatment intensity: (1) inpatient treatment program (5 days a week), (2) day treatment program (4 days a week), and (3) a part-time outpatient treatment program of two half days per week. Patients attend one of these programs and stay in the program for at least 6 months (with an average duration of 8 months). For pragmatic reasons, patients are not randomized across the treatment programs. Sensitivity analyses will be performed and if appropriate given our sample size, differences in baseline characteristics and treatment effects between the programs will be investigated.

Self-report questionnaires on personality functioning, symptoms, resilience, quality of life, epistemic trust, mentalizing and the therapeutic alliance are filled out via REDCAP, an online platform, at baseline, after 3 and 6 months of treatment, at discharge, and 6-months and at 1 and 2 year follow-up. Automated invitations and reminders are sent via e-mail. Automated scoring and codebooks are implemented via REDCAP. A designated study data manager follows up participant progress and provides support. The data manager additionally logs drop-out including the reason for treatment termination and the occurrence of the following serious adverse events (SAE's): suicide attempt, life-threatening self-harm, patient death, serious injury or medical disease that requires hospitalization.

References:

American Psychiatric Association. (2013). Diagnositic and statistical manual of mental disorders (5th ed.). Arlington, VA: American Psychiatric Publishing. https://doi.org/10.1176/appi.books.9780890425596.744053

Budge, S. L., Moore, J. T., Del Re, A. C., Wampold, B. E., Baardseth, T. P., & Nienhuis, J. B. (2013). The effectiveness of evidence-based treatments for personality disorders when comparing treatment-as-usual and bona fide treatments. Clin Psychol Rev, 33(8), 1057-1066. https://doi.org/10.1016/j.cpr.2013.08.003

Cristea, I. A., Gentili, C., Cotet, C. D., Palomba, D., Barbui, C., & Cuijpers, P. (2017). Efficacy of Psychotherapies for Borderline Personality Disorder: A Systematic Review and Meta-analysis. Jama Psychiatry, 74(4), 319-328. https://doi.org/10.1001/jamapsychiatry.2016.4287

Fonagy, P., Luyten, P., Allison, E., & Campbell, C. (2019). Mentalizing, Epistemic Trust and the Phenomenology of Psychotherapy. Psychopathology. https://doi.org/10.1159/000501526

Grant, B. F., Chou, S. P., Goldstein, R. B., Huang, B., Stinson, F. S., Saha, T. D., Smith, S. M., Dawson, D. A., Pulay, A. J., Pickering, R. P., & Ruan, W. J. (2008). Prevalence, correlates, disability, and comorbidity of DSM-IV borderline personality disorder: results from the Wave 2 National Epidemiologic Survey on Alcohol and Related Conditions. Journal of Clinical Psychiatry, 69(4), 533-545. https://doi.org/10.4088/jcp.v69n0404

Gregory, R. J., & Sachdeva, S. (2016). Naturalistic Outcomes of Evidence-Based Therapies for Borderline Personality Disorder at a Medical University Clinic. Am J Psychother, 70(2), 167-184. https://doi.org/10.1176/appi.psychotherapy.2016.70.2.167

Jacobson, N. S., & Truax, P. (1991). Clinical significance: a statistical approach to defining meaningful change in psychotherapy research. J Consult Clin Psychol, 59(1), 12-19. https://doi.org/10.1037//0022-006x.59.1.12

Kramer, U. (2018). Mechanisms of Change in Treatments of Personality Disorders: Introduction to the Special Section. Journal of Personality Disorders, 32(Suppl), 1-11. https://doi.org/10.1521/pedi.2018.32.supp.1

Lowyck, B., Vermote, R., Verhaest, Y., Vandeneede, B., Wampers, M., Luyten, P., & Wampers, M. (2015). Hospitalization-based psychodynamic treatment for personality disorders: A five-year follow-up. Psychoanalytic Psychology, 32, 381-402. https://doi.org/10.1037/a0038959

MacCallum, R. C., Kim, C., Malarkey, W. B., & Kiecolt-Glaser, J. K. (1997). Studying multivariate change using multilevel models and latent curve models. Multivariate Behavioral Research, 32, 215-253. https://doi.org/10.1207/s15327906mbr3203

Malmivaara, A. (2015). Benchmarking Controlled Trial--a novel concept covering all observational effectiveness studies. Ann Med, 47(4), 332-340. https://doi.org/10.3109/07853890.2015.1027255

Storebø, O. J., Stoffers-Winterling, J. M., Völlm, B. A., Kongerslev, M. T., Mattivi, J. T., Jørgensen, M. S., Faltinsen, E., Todorovac, A., Sales, C. P., Callesen, H. E., Lieb, K., & Simonsen, E. (2020). Psychological therapies for people with borderline personality disorder. Cochrane Database Syst Rev, 5(5), Cd012955. https://doi.org/10.1002/14651858.CD012955.pub2

Winsper, C., Bilgin, A., Thompson, A., Marwaha, S., Chanen, A. M., Singh, S. P., Wang, A., & Furtado, V. (2020). The prevalence of personality disorders in the community: a global systematic review and meta-analysis. The British Journal of Psychiatry, 216(2), 69-78. https://doi.org/10.1192/bjp.2019.166

ELIGIBILITY:
Inclusion Criteria:

1. Individuals (male, female, non-binary or other) older than 18 years
2. Meeting criteria for personality disorder as assessed by a psychiatrist and confirmed with the PID-5 and LFPS self-report scales
3. Sufficient mastery of the Dutch language to follow treatment and complete questionnaires
4. Agreeing to participate in the study following informed consent procedure

Exclusion Criteria:

1. Substance abuse that would interfere with the ability to adhere to the treatment
2. Acute psychotic symptoms as assessed by a psychiatrist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be consecutively admitted patients to the Klipp treatment unit at the University Psychiatric Center (UPC) KU Leuven, Campus Kortenberg (Belgium) which provides specialized treatment for PDs, starting from April 17 2023 until the target sample size of N = 110 is reached.
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2026-04-17 (Estimated); Study Completion 2028-04-17 (Estimated)

PRIMARY OUTCOMES:
Changes in General Psychological Symptoms | From baseline to treatment termination (on average 9 months after the start of treatment)
  Self-reported severity of general psychological symptoms as assessed using the Brief Symptom Inventory (BSI; Derogatis & Melisaratos, 1983).

SECONDARY OUTCOMES:
Changes in Borderline Personality Disorder Symptom Severity | From baseline to treatment termination (on average 9 months after the start of treatment), and at 6-month, and one- and two-year follow-up
  Self-reported severity of borderline symptomatology and assessed via the Personality Assessment Inventory - Borderline subscale (PAI-BOR; Distel et al. (2009)).
Changes in General Psychological Symptoms | From baseline to 6-month, and one- and two-year follow-up
  Self-reported severity of general psychological symptoms as assessed using the Brief Symptom Inventory (BSI; Derogatis & Melisaratos, 1983).
Changes in Personality Functioning | From baseline to treatment termination (on average 9 months after the start of treatment), and 6-month, and one- and two-year follow-up
  Self-reported severity of personality pathology, as measured using the Level of Personality Functioning Scale (LPFS; Hutsebaut et al., 2015)
Changes in Interpersonal Problems | From baseline to treatment termination (on average 9 months after the start of treatment), and 6-month, and one- and two-year follow-up
  Self-reported severity of interpersonal problems assessed with the Inventory of Interpersonal Problems (IIP; Barkham et al., 1996)
Changes in Symptoms of Post-traumatic Stress | From baseline to treatment termination (on average 9 months after the start of treatment), and 6-month, and one- and two-year follow-up
  Self-reported severity of symptoms of Post-traumatic Stress Disorder (PTSD), assessed with the PTSD Checklist for DSM-5 (PCL-5; Van Praag et al., 2020)
Changes in Resilience | From baseline to treatment termination (on average 9 months after the start of treatment), and 6-month, and one- and two-year follow-up
  Self-reported resilience to deal with life stressors, measured with the Connor-Davidson Resilience Scale (CD-RISC; Connor & Davidson, 2003)
Changes in Quality of Life | From baseline to treatment termination (on average 9 months after the start of treatment), and 6-month, and one- and two-year follow-up
  Self-reported health-related quality of life as assessed with the EuroQol Quality of life 5 dimensions (EQ-5D; Herdman et al., 2011)

OTHER OUTCOMES:
Change Mechanisms | At baseline, after 3 months of treatment, 6 months of treatment and at treatment termination (on average 9 months after the start of treatment)
  We will investigate whether change trajectories across treatment in epistemic trust (Epistemic Trust, Mistrust and Credulity Questionnaire; ETMCQ) are associated with symptom change trajectories across treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Celine De Meulemeester, PhD, Principal Investigator — KU Leuven
Locations (1):
- University Psychiatric Center KU Leuven, Kortenberg, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Yes
IPD will be made available upon reasonable request from other researchers, including a research plan of how they plan to use the data.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: After publication of the study's main results.
Access Criteria: Requests can be made by other researchers by contacting the corresponding author of the study publications via e-mail. The requests will be evaluated by the Prinicipal Investigator. IPD will be made available for meta-analyses or other follow-up studies. De-identified data will be shared via the secure data transfer application Send-it in REDCAP. The recipient will receive an email containing a unique download URL, along with a second follow-up email with the password (for greater security) for downloading the file. The file will be stored securely and then later removed from the server after the specified expiration date.